CLINICAL TRIAL: NCT05926466
Title: A Phase IIb, Open-Label, Randomized Controlled Dose Ranging Multi-Center Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Exposure-Response Relationship of Different Doses of BTZ-043 in Combination With Bedaquiline and Delamanid in Adult Subjects With Newly Diagnosed, Uncomplicated, Drug-sensitive Pulmonary Tuberculosis
Brief Title: BTZ-043 Dose Evaluation in Combination and Selection
Acronym: DECISION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Hoelscher (Other)
Collaborators: Radboud University Medical Center (Other); University of California, San Francisco (Other); University College, London (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Director, Division for Infectious Diseases and Tropical Medicine, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMU-IMPH-BTZ-043-04; UNITE4TB-02 (Other: UNITE4TB)
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Tuberculosis, Pulmonary; Other Specified Pulmonary Tuberculosis
Keywords: Tuberculosis; BTZ-043; Bedaquiline; Delamanid; Moxifloxacin; Safety; Tolerability; Pharmacokinetics (PK); Benzothiazinones; Pulmonary Tuberculosis; Dose-finding; Antitubercular agents
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — 2-(2-methyl-1,4-dioxa-8-azaspiro(4.5)dec-8-yl)-8-nitro-6-(trifluoromethyl)-4H-1,3-benzothiazin-4-one; bedaquiline; OPC-67683; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: The study will compare the efficacy, safety of 3 experimental regimens with a comparator regimen administered over 16 weeks, in participants with newly diagnosed, drug sensitive pulmonary tuberculosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Active Comparator): Drug: Moxifloxacin Moxifloxacin will be dosed at the licensed dose of 400 mg orally once daily for 16 weeks Drug: Bedaquiline Bedaquiline will be dosed at 400 mg orally once daily for the first 2 weeks, followed by 100 mg orally once daily for 14 weeks Drug: Delamanid Delamanid will be dosed at 300 mg orally once daily for 16 weeks
  Interventions: Drug: Bedaquiline; Drug: Delamanid; Drug: Moxifloxacin
- Arm 2 (Experimental): Drug: Bedaquiline Bedaquiline will be dosed at 400 mg orally once daily for the first 2 weeks, followed by 100 mg orally once daily for 14 weeks Drug: Delamanid Delamanid will be dosed at 300 mg orally once daily for 16 weeks Drug: BTZ-043 BTZ-043 will be dosed at 500 mg orally once daily for 16 weeks
  Interventions: Drug: BTZ-043; Drug: Bedaquiline; Drug: Delamanid
- Arm 3 (Experimental): Drug: Bedaquiline Bedaquiline will be dosed at 400 mg orally once daily for the first 2 weeks, followed by 100 mg orally once daily for 14 weeks Drug: Delamanid Delamanid will be dosed at 300 mg orally once daily for 16 weeks Drug: BTZ-043 BTZ-043 will be dosed at 1000 mg orally once daily for 16 weeks
  Interventions: Drug: BTZ-043; Drug: Bedaquiline; Drug: Delamanid
- Arm 4 (Experimental): Drug: Bedaquiline Bedaquiline will be dosed at 400 mg orally once daily for the first 2 weeks, followed by 100 mg orally once daily for 14 weeks Drug: Delamanid Delamanid will be dosed at 300 mg orally once daily for 16 weeks Drug: BTZ-043 BTZ-043 will be dosed at 1500 mg orally once daily for 16 weeks
  Interventions: Drug: BTZ-043; Drug: Bedaquiline; Drug: Delamanid

INTERVENTIONS:
Drug: BTZ-043 — BTZ-043 belongs to the chemical class of benzothiazinones, and is a promising antibiotic for the treatment of Tuberculosis. Its mechanism of action is based on the covalent inhibition of the enzyme decaprenylphosphoryl-ß-D-ribose-2'-epimerase (DprE1), which is essential for the cell wall assembly of mycobacteria. . Formation of the covalent adduct between BTZ-043 and DprE1 results in inhibition of cell wall biosynthesis and loss of viability of Mycobacteria Tuberculosis. BTZ-043 has been evaluated in three clinical studies: a phase Ia, First Time in Human study (FTIH), a two-stage phase Ib multiple ascending dose (MAD) and phase IIa monotherapy early bactericidal activity (EBA) study, and a human ADME (Absorption/Distribution/Metabolism/Excretion) study.
  Arms: Arm 2; Arm 3; Arm 4
Drug: Bedaquiline — Bedaquiline, is a diarylquinoline compound with a novel mechanism of action against MTB, the inhibition of mycobacterial adenosine triphosphate (ATP) synthase. On the 28th of December 2012, the Food and Drug Administration (FDA) granted accelerated approval to SIRTURO® (bedaquiline) tablets as a part of combination therapy in adults with MDR-TB. It is the first to be introduced specifically for the treatment of MDR-TB in combination with other drugs.
  Other Names: SIRTURO®
Drug: Delamanid — Delamanid is a nitro-dihydro-imidazooxazole derivative that inhibits the synthesis of mycolic acids, a crucial component of the cell wall of MTB. Delamanid has received regulatory approvals in several countries and is currently recommended by WHO for for use in longer MDR- or RR-TB regimens in line with WHO recommendations.
  Other Names: OPC-67683; Deltyba
Drug: Moxifloxacin — Moxifloxacin belongs to the group of fluoroquinolones (FQ). FQs are a mainstay of MDR-TB treatment, and Moxifloxacin is considered the most potent drug in second line MDR-TB therapy, recently reviewed by WHO, with only moderate pre-existing resistance in the community.
  Other Names: Lonxave
  Arms: Arm 1

SUMMARY:
This is a phase 2B, open label study, that will compare the safety and efficacy of three experimental regimens consisting of bedaquiline and delamanid in combination with different doses of BTZ-043, a novel antibiotic, in adult participants with newly diagnosed, drug-sensitive pulmonary tuberculosis. Participants will be assigned to receive either one of the three BTZ-043-containing regimens or a comparator regimen consisting of bedaquiline, delamanid and moxifloxacin. The objective is to find the optimal dose of BTZ-043 with the highest efficacy and safety to be used in subsequent studies.

DETAILED DESCRIPTION:
This open label, phase 2B, randomized controlled study will evaluate three experimental arms containing different doses of BTZ-043 in combination with bedaquiline and delamanid, in adult subjects with newly diagnosed, drug-sensitive pulmonary tuberculosis, in comparison with bedaquiline, delamanid and moxifloxacin, administered over 16 weeks. A total of 90 adult (≥ 18 years of age) participants will be enrolled. In case of a high number of dropouts or non-evaluable participants, it may be necessary to recruit more participants into the study.

The participants will be randomly allocated to one of the three BTZ-containing experimental regimens or the moxifloxacin-containing comparator regimen:

Arm 1: bedaquiline, delamanid, BTZ-043 500 mg (BDT500) Arm 2: bedaquiline, delamanid, BTZ-043 1000 mg (BDT1000) Arm 3: bedaquiline, delamanid, BTZ-043 1500 mg (BDT1500) Arm 4: bedaquiline, delamanid, moxifloxacin (BDM) In all arms, bedaquiline will be dosed at 400 mg once daily for 2 weeks, followed by 100 mg once daily for 14 weeks and delamanid will be dosed at 300 mg once daily for 16 weeks. Moxifloxacin will be dosed at 400 mg once daily in the comparator arm. After completion of 16 weeks of treatment, all participants will receive 8 weeks of continuation therapy with Rifampicin and Isoniazid.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures, including HIV testing.
* Male or female, aged 18 up to (and including) 64 years.
* Body weight (in light clothing and with no shoes) within the range of 30 to 100kg and body mass index within the range of 15 to 40kg/m2.
* Newly diagnosed, previously untreated current episode of drug-susceptible pulmonary TB (presence of MTB complex with rapid molecular test result confirming susceptibility to rifampicin and isoniazid such as "GeneXpert" and/or "HAIN MTBDR plus").
* ≥ 1 sputum sample from concentrated spot sputum positive in GeneXpert MTB/RIF Ultra®, with semi-quantitative result at least "medium" or higher.
* FEMALE PARTICIPANTS: Inability to conceive AND/OR inability of partner(s) to father children OR consent to use effective methods of contraception when engaging in heterosexual intercourse, as defined below:

  a. Non-childbearing potential: i) Bilateral oophorectomy AND/OR hysterectomy OR bilateral tubal ligation more than 12 months ago, AND/OR has been postmenopausal with a history of no menses for at least 12 consecutive months as per medical history.

ii) Sexual partner(s) of female participant: vasectomy OR bilateral orchidectomy at least three months prior to screening as per medical history.

b. Effective contraception methods: i) Two methods, including methods used by patient's sexual partner(s). At least one must be a barrier method. Contraception must be practised for at least until 12 weeks after the last dose of BTZ-043.

- MALE PARTICIPANTS: Inability to father children AND/OR inability of partner(s) to conceive, OR consent to use effective methods of contraception when engaging in heterosexual intercourse, as defined below:

c. Non-childbearing potential: i) Sexual partner(s) of male participant: Bilateral oophorectomy AND/OR hysterectomy OR bilateral tubal ligation more than 12 months ago, AND/OR has been postmenopausal with a history of no menses for at least 12 consecutive months as per medical history.

ii) Vasectomy OR bilateral orchidectomy at least three months prior to screening as per medical history.

iii) Female pregnant sexual partner of a male participant: agree to use at least one barrier method.

iv) Male sexual partner of male participant: agree to use at least one barrier method for at least until 12 weeks after the last dose of BTZ-043 for protection of the partner.

d. Effective contraception methods: ii) Two methods, including methods used by patient's female sexual partner(s). At least one must be a barrier method. Effective contraception must be ensured for at least 16 weeks after the last dose of BTZ-043

Exclusion Criteria:

* Circumstances that raise doubt about free, unconstrained consent to study participation (e.g. in a prisoner or person suffering from an intellectual disability).
* Poor general condition, where delay in treatment cannot be tolerated, or death within three months is likely, as assessed by the investigator.
* Poor social condition which would result in a high likelihood of not completing the trial until the final visit.
* The patient is pregnant or breast-feeding.
* The patient is HIV antibody positive (known, or on a test performed at screening), unless:

  1. The patient has a viral load (VL) < 200 copies/mL on a test performed at screening
  2. The patient has a CD4 cell count > 200 cells/mm3 at screening
  3. The patient is experienced on antiretroviral therapy (ART), and is on a combination of tenofovir, lamivudine and dolutegravir (TDF/3TC/DTG) for a minimum of 6 months prior to the screening visit.
* The patient has a known intolerance to any of the study drugs or concomitant disorders or conditions for which study drugs or standard TB treatment are contraindicated.
* The patient has received treatment with any other investigational drug within 1 month prior to enrolment, or is planning to be enrolled into other clinical (intervention) trials during participation.
* The patient has a history of or current evidence of clinically relevant cardiovascular, metabolic, gastrointestinal, neurological, ophthalmological, psychiatric or endocrine diseases, malignancy or any other condition, that will influence treatment response, study adherence or survival in the judgement of the investigator, especially:

  1. Clinically significant evidence of severe or extra-thoracic TB (e.g., miliary TB, TB meningitis, excluding limited lymph node involvement)
  2. Serious lung conditions other than TB or significant respiratory impairment in the discretion of the investigator
  3. Peripheral neuropathy (as evaluated by the Brief Peripheral Neuropathy Score).
  4. Significant psychiatric disorder like depression or schizophrenia; especially if treatment for those has ever been required in the last five years or is anticipated to be required.
  5. An established diagnosis of diabetes mellitus.
  6. Cardiovascular disease, such as myocardial infarction, heart failure, coronary heartdisease, arrhythmia, tachyarrhythmia, or pulmonary hypertension.
  7. Current (as measured on two occasions during screening) or history of hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure of ≥90 mmHg) on two occasions. Controlled hypertension is permitted if the patients receive only the allowed anti-hypertensives.
  8. Long QT syndrome or family history of long QT syndrome or sudden death of unknown or cardiac-related cause.
  9. Alcohol or other drug abuse, that is sufficient to significantly compromise the safety or cooperation of the patient, includes substances prohibited by the protocol, or has led to significant organ damage, at the discretion of the investigator. An isolated positive test for cannabinoids does not fulfil this exclusion criterion.
  10. Chronic kidney disease (CKD) or any other history of renal impairment.
* Any of the following laboratory findings at screening:

  1. serum amino aspartate transferase (AST) and/or alanine aminotransferase (ALT) activity >3x the ULN
  2. serum alkaline phosphatase (ALP) >3x the ULN
  3. serum total bilirubin level >1.5 times the ULN
  4. estimated creatinine clearance (eCrCl) < 60 mls/min (calculated using the Cockcroft and Gault formula
  5. haemoglobin level <8.0 g/dL
  6. platelet count <50,000/mm3
  7. albumin < 2.8 g/dl
  8. serum potassium <3.5 mmol/L (not excluded if subsequently corrected)
  9. serum magnesium < 0.5mmol/L (not excluded if subsequently corrected)
* Any of the following ECG findings at screening:

  1. QTcF of > 450 milliseconds (ms)
  2. Atrioventricular (AV) block with PR interval > 200 ms
  3. QRS complex > 120 ms
  4. any other changes in the ECG that are clinically relevant as per discretion of the investigator
* Any of the following regarding concomitant medications at screening:

  1. Previous treatment with first- and second-line anti-TB drugs within the last 3 months prior to screening.
  2. Treatment with any other investigational drug (including vaccines) within 1 month prior to enrolment or enrolment into other clinical (interventional) trials during participation.
  3. Unable or unwilling to only take the allowed concomitant medications for this studyand ensuring an appropriate washout period
  4. Unable or unwilling to abide to the dietary restrictions required in this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Time to positivity in BD MGIT liquid culture | Day 01- Day 112
  To evaluate which of the BTZ-043 containing experimental arms is superior, the change in mycobacterial load over time on treatment as quantified by time to positivity in BD MGIT 960® (Mycobacterium Growth Tube Indicator) liquid culture described by non-linear mixed-effects methodology

SECONDARY OUTCOMES:
Time to stable culture conversion to negative in liquid media | Day 01- Day 112
  The time on treatment required until a participant achieves the first of two successive visits with negative cultures without an intervening positive culture
Proportion of participants converting to negative sputum culture in liquid media | Day 01- Day 112
  Proportion of participants converting to negative sputum culture in liquid media defined as two consecutive negative cultures without an intervening positive culture) at each time point during treatment
Frequency of all adverse events (serious and non-serious) | Day 01- Day 168
  To assess the frequency, severity, and type of adverse events (AEs), and AE related treatment discontinuations.
Frequency of adverse events of Grade 3 severity (severe) or higher | Day 01- Day 168
  Severity of AEs will be classified following the U.S. National Institutes of Health Common Terminology Criteria for Adverse Events 5.0 (CTCAE). The minimum grade is 1 (Mild) and the maximum grade is 5 (Death related to AE).
  Higher scores mean a worse outcome
Frequency of adverse events possibly, probably or definitely related to study drug | Day 01- Day 168
  To assess the frequency, severity, and type of adverse events (AEs), and AE related treatment discontinuations.
Frequency of treatment discontinuations or interruptions related to adverse events/serious adverse event | Day 01- Day 168
  To assess the frequency, severity, and type of adverse events (AEs), and AE related treatment discontinuations.
Changes in ECG intervals of PR, RR, QRS, QT, Fridericia-corrected QT [QTcF] | Day 01- Day 168
  • Proportion of participants with QTcF > 500ms in ECGs on treatment. • Proportion of participants who have a QTcF prolongation of grade 3 or higher
Area under the plasma concentration curve from dosing to the end of the dosing interval (AUC 0-24) | Day 28, Day 56
  The pharmacokinetics parameters will be assessed for BTZ-043, bedaquiline and delamanid, and their major metabolites (Arm 2-4), in all participants. Extensive sampling will be done for BTZ-043 at the WK04 visit (Day 28 ± 2 Days) and sparse PK sampling for bedaquiline and delamanid on WK04 (Day 28 ± 2 Days) and WK08 visits (Day 56 ± 2 Days)
The observed maximum concentration (Cmax) | Day 28, Day 56
  The pharmacokinetics parameters will be assessed for BTZ-043, bedaquiline and delamanid, and their major metabolites (Arm 2-4), in all participants. Extensive sampling will be done for BTZ-043 at the WK04 visit (Day 28 ± 2 Days) and sparse PK sampling for bedaquiline and delamanid on WK04 (Day 28 ± 2 Days) and WK08 visits (Day 56 ± 2 Days)
Time to reach Cmax (Tmax) | Day 28, Day 56
  The pharmacokinetics parameters will be assessed for BTZ-043, bedaquiline and delamanid, and their major metabolites (Arm 2-4), in all participants. Extensive sampling will be done for BTZ-043 at the WK04 visit (Day 28 ± 2 Days) and sparse PK sampling for bedaquiline and delamanid on WK04 (Day 28 ± 2 Days) and WK08 visits (Day 56 ± 2 Days)
Minimum observed plasma concentration 24 hours following the last dose (Cmin) | Day 28, Day 56
  The pharmacokinetics parameters will be assessed for BTZ-043, bedaquiline and delamanid, and their major metabolites (Arm 2-4), in all participants. Extensive sampling will be done for BTZ-043 at the WK04 visit (Day 28 ± 2 Days) and sparse PK sampling for bedaquiline and delamanid on WK04 (Day 28 ± 2 Days) and WK08 visits (Day 56 ± 2 Days)
Apparent oral clearance (Cl/F) | Day 28, Day 56
  The pharmacokinetics parameters will be assessed for BTZ-043, bedaquiline and delamanid, and their major metabolites (Arm 2-4), in all participants. Extensive sampling will be done for BTZ-043 at the WK04 visit (Day 28 ± 2 Days) and sparse PK sampling for bedaquiline and delamanid on WK04 (Day 28 ± 2 Days) and WK08 visits (Day 56 ± 2 Days)
Terminal half-life (t 1/2) | Day 28, Day 56
  The pharmacokinetics parameters will be assessed for BTZ-043, bedaquiline and delamanid, and their major metabolites (Arm 2-4), in all participants. Extensive sampling will be done for BTZ-043 at the WK04 visit (Day 28 ± 2 Days) and sparse PK sampling for bedaquiline and delamanid on WK04 (Day 28 ± 2 Days) and WK08 visits (Day 56 ± 2 Days)
Identification of M. tuberculosis complex and Isoniazid (INH) resistance by PCR (GeneXpert Ultra MTB/RIF®/ GeneXpert XDR/HAIN MTBDRplus or similar) | Day 01-Day 112
  Cultures grown from the screening period, and the last sputum sample with mycobacteriological growth will be assessed. This test is qualitative, therefore the result will be: Detected, not detected or indeterminate
Minimum inhibitory concentrations (MIC) of study drugs the patient was receiving | Day 01- Day 112
  Cultures grown from the screening period, and the last sputum sample with mycobacteriological growth will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Prof Dr, Study Director — LMU University Hospital
Locations (4):
- South Africa (2):
  - TASK Applied Sciences Clinical Research Centre, Cape Town
  - TASK Applied Science Eden, George
- Tanzania (2):
  - National Institute for Medical Research (NIMR-MMRC), Mbeya
  - National Institute for Medical Research (NIMR-Mwanza),, Mwanza